CLINICAL TRIAL: NCT00639457
Title: Exercise and Pioglitazone for HIV-Metabolic Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kevin Yarasheski, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK 049393 (completed); WU 157 (Other: ACTU Washington University)
Record Dates: First submitted 2008-03-18; First posted 2008-03-20 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Type 2 Diabetes; Obesity; HIV; AIDS; Cardiovascular Disease; Lipodystrophy
Keywords: PPAR-gamma agonist; glucose metabolism; inflammation; adipose tissue distribution; cardiac function; vascular function; mass spectrometry; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Diabetes Mellitus, Type 2; Obesity; Acquired Immunodeficiency Syndrome; Cardiovascular Diseases; Lipodystrophy; Inflammation | interventions — Pioglitazone; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone (Actos; 30mg/day) for 16 weeks.
  Interventions: Drug: Pioglitazone
- Pioglitazone + Exercise training (Active Comparator): Pioglitazone (Actos; 30mg/day) plus progressive aerobic and weight lifting exercise training (1.5hr/day x 3 days/wk)supervised and monitored by a personal exercise trainer.
  Interventions: Drug: Pioglitazone; Behavioral: Exercise training

INTERVENTIONS:
Drug: Pioglitazone — Oral 30mg/day for 16 weeks
  Other Names: Actos
Behavioral: Exercise training — Supervised aerobic and resistance exercise training (1.5hrs/day x 3 days/wk) for 16 weeks
  Other Names: Physical activity
  Arms: Pioglitazone + Exercise training

SUMMARY:
The purpose is to examine the safety and efficacy of 16wks of pioglitazone (Actos; 30mg/d) with and without aerobic and strength exercise training for reducing glucose intolerance and central adiposity in HIV-infected people. We anticipate that pioglitazone + exercise training will improve glucose metabolism and insulin sensitivity, and reduce central adiposity more than pioglitazone alone. These improvements should translate into reduced cardiovascular disease risk in HIV-infected people.

DETAILED DESCRIPTION:
Our prior research has examined the pathogenesis and potential treatments for metabolic complications in people living with HIV. We have adopted the "lipotoxicity" hypothesis for Metabolic Syndrome X to explain the pathogenesis of impaired glucose tolerance (IGT) and fat redistribution in HIV: increased lipolysis and mobilization of lipids and free fatty acids from subcutaneous adipose depots leads to their excessive deposition in muscle and liver which contributes to dyslipidemia, insulin resistance, increased hepatic glucose output, and possibly visceral fat accumulation. Effective treatments have not been identified. Consensus groups recommend regular exercise and dietary modifications as primary and pharmacologic interventions as secondary treatments for the syndromes. We propose to test the efficacy of aerobic and weight lifting exercise training and an oral insulin-sensitizing agent (pioglitazone) as treatments for HIV-associated IGT and fat redistribution. We propose a 4-month, 2-group randomized study to evaluate the efficacy of pioglitazone and exercise + pioglitazone in 40 men and 40 women living with HIV and IGT and fat redistribution. We will measure: insulin sensitivity, glucose disposal rate, hepatic glucose production rate (5hr-hyperinsulinemic euglycemic clamp with 6,6-[2H2]-glucose); whole-body and regional fat and muscle content (1H-MRI of the abdomen and thigh & DEXA), soleus muscle and liver lipid content (1H-MRS), muscle and fat PPARgamma/alpha mRNA and protein expression, serum lipid profiles, and serum adiponectin levels before and at the end of 4 months of treatment. We hypothesize that exercise training + pioglitazone will be more effective than pioglitazone alone at improving insulin sensitivity, reducing visceral fat, liver and muscle lipid content, and increasing peripheral subcutaneous fat content in HIV-infected people. We hypothesize that combined treatment will be more effective because exercise training will activate PPARalpha expression in muscle and pioglitazone will activate PPARy expression in fat and muscle. We anticipate that this project will provide direct evidence that supports the combined use of exercise training and pioglitazone in people living with HIV and experiencing metabolic and anthropomorphic disorders that increase cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 yr old HIV-infected men (n=40) and women (n=40).
2. Source documentation of HIV status.
3. Stable on highly active antiretroviral therapy (HAART) that may or may not include HIV-protease inhibitors for at least 3 months prior to enrollment. As of Jan 2005, HIV-infected long-term non-progressors will be included, even though they are not receiving HAART because it is likely that their disease status will not advance during the study period.
4. Impaired glucose tolerance (IGT) or type 2 diabetes and fat redistribution. IGT is defined as: fasting (8hr) plasma glucose 100-126mg/dL or plasma glucose >140 mg/dL 2-hours after a 75g-oral glucose load. This definition (proposed/revised May 2006) includes volunteers with adult onset type 2 diabetes (non-insulin dependent diabetes), because we believe that these volunteers may benefit from the potential glucose-lowering actions of pioglitazone with or without exercise training. Fat redistribution is defined as any 2 of the following: waist-to-hip ratio >0.85 women or >0.95 men, or trunk/appendicular adipose ratio using whole-body DEXA >0.85 women or >1.3 men, or <15% leg fat (DEXA; (leg fat/total body fat) x100), or visceral adiposity VAT >120 cm2 women or >140 cm2 men, or a VAT/TAT ratio >0.30 women or >0.40 men. Overall, the eligibility criteria are designed to include subjects with metabolic syndromes that increase CVD risk, and the potential to gain the greatest benefit from pioglitazone and exercise training. These inclusion criteria will help select/maintain homogeneous groups of study participants.
5. Plasma HIV RNA (Roche Amplicor® assay) <5000 copies/ml OR a CD4 T-cell count >100 cells/µL and stable for previous 3 months.
6. BMI 20-40kg/m2.
7. "Normal" blood chemistries for at least 1 month prior to enrollment; platelet count >30,000/mm3, absolute neutrophil count <750/mm3, transaminases <2.5x the upper limit of normal (ULN), creatinine <3x ULN, fasting triglycerides <500 mg/dL.

Exclusion Criteria:

1. Medications or agents that might alter/impair glucose metabolism (insulin, glucocorticoids, corticosteroids, megace) during the 3 months prior to enrollment or at any time during enrollment. Volunteers who developed type 2 diabetes after HIV-infection or after starting anti-HIV medications, who are receiving insulin sensitizers (metformin, meglitinides, alpha-glucosidase inhibitors) or insulin secretagogues (sulfonylureas), but still do not have their blood sugars in control (defined as IGT above) are eligible.
2. Abnormal or unstable (for 3 months prior to enrollment) endocrine blood chemistries that might otherwise explain insulin resistance. TSH <0.2 or >12µIU/mL, morning cortisol >22µg/dL, IGF-1 <115ng/mL, total testosterone <200ng/dL (men) <15ng/dL (women). Use of testosterone, ACTH, thyroid hormone, or rhGH replacement to normalize low levels is permitted, but must be stable on hormone replacement for 3 months prior to enrollment and will not discontinue this replacement during enrollment. Hormone replacement cannot be started during treatment.
3. Allergy or hypersensitivity to thiazolidinediones. Currently taking a thiazolidinedione.
4. Anti-obesity or anorectic medications during the 3 months prior to enrollment or at any time during enrollment. Lipid-lowering medications are permitted (fibrate or statin), but the subject must be stable on that agent for at least 3 months prior to enrollment. Lipid-lowering agents cannot be started during the treatment period.
5. Chronic hepatitis B infection (HB surface antigen positive). Active hepatitis C infection (detectable Hep C RNA). Those who have cleared hepatitis B or C infection are eligible. This was revised in May 2006 to better clarify some uncertainties about hepatitis and eligibility.
6. History of serious cardiovascular conditions or NY Heart Association (NYHA) cardiac status Class III or IV, (e.g., recent MI, unstable angina, edema, CHF, CAD, CABG, valve disease (murmur), stroke, uncontrolled high blood pressure (resting >140/90 mmHg on 3 occasions), irregular heart rhythm, bundle-branch block, aortic stenosis, resting ST-segment depression >1mm) that would preclude exercise testing/training, or substantially increase risk of a CV-event during exercise, or would limit the subjects ability to participate in exercise training. Treatment with medications for a cardiovascular condition (cardiac glycosides, alpha- or beta-blockers). Some antihypertensive medications (Ca++-channel blocker, diuretic, or ACE inhibitor) will be permitted.
7. Insulin-dependent diabetes mellitus (IDDM) or a history of ketoacidosis, symptomatic diabetic neuropathy or retinopathy, or renal disease (creatinine >3x ULN).
8. Hematocrit <34% in men or <25% in women with symptoms (fatigue, "tired-legs", shortness of breath). Hemoglobin <10 gm/100ml with symptoms.
9. History of eating disorder, significant GI-disease
10. Nausea, vomiting, diarrhea (>4 loose stools/day) that are unresponsive to treatment during 2wks prior to enrollment or that persists for >2wks during enrollment.
11. Active secondary infection. Any significant change in chronic suppressive therapy for an opportunistic infection during the 1-month prior to enrollment.
12. During the 3 months prior to enrollment, regular aerobic or weight lifting exercise training that exceeds the minimum (45min/d, 3d/wk, >75% exercise capacity) required for the metabolic, biochemical, and anthropomorphic benefits of exercise to be attained as described in the American College of Sports Medicine Guidelines. In Apr 2006, this exclusion criterion was modified in order to facilitate enrollment of volunteers who are moderately-highly active during the 3months prior to screening for this study. We will randomize volunteers who exercise regularly into the two treatment groups. This will reduce the potential confounding effects of regular exercise on the metabolic, biochemical, and anthropomorphic benefits of exercise training that is prescribed during the treatment phase. We have excluded several volunteers who are regular exercisers, and we believe we may be unnecessarily excluding them. They can be included, enrollment will be facilitated, and the study design will not be adversely affected, as long as we randomize them into pioglitazone or exercise+pioglitazone (1:1).
13. Unwilling or unable to do supervised exercise 3 sessions/wk at the Medical School exercise facility. Any condition that might be contraindicated for exercise training (disabling joint, cartilage or muscle injury/disorder that prohibits or severely limits participation in regular exercise, disabling arthritis, severe physical disabilities, claudication, pulmonary disease, sinus tachycardia, arrhythmias, premature atrial or ventricular contractions).
14. Pregnancy or nursing mothers. Women cannot be pregnant and must agree to use an acceptable form of birth control during the treatment period. If birth control pills are used, the woman must be stable on these medications for at least 6 months prior to enrollment. All metabolic testing will be done in the early follicular phase. Urine pregnancy tests (hCG) will be done at baseline and every month the woman is enrolled in the study.
15. Pancreatitis within prior 1 year. Serum triglycerides >500mg/dL esp. with history of pancreatitis, or otherwise at high risk for pancreatitis.
16. Medications that inhibit or slow blood coagulation (ie., blood thinners). Prothrombin (clotting) time exceeds 2 sec > control (only in subjects who agree to muscle/fat biopsies).
17. Active malignancy or treatment with chemotherapeutic agents or radiation therapy during the 3 months prior to enrollment.
18. Excessive weight loss (>10% body weight) during the 3 months prior to enrollment. History of hyperlactatemia or lactic acidosis, esp. with rapid weight loss.
19. "Blinded" investigational drugs/medications during the 3 months prior to enrollment that will not be unblinded before enrollment. Open-label investigational drugs are permitted. Must be stable on these for 3 months prior to enrollment, must remain stable on them during the treatment period, and they must be known not to affect glucose, lipid, adipose tissue or liver metabolism.
20. Non-prescription over the counter drugs/supplements that might alter glucose, lipid, or adipose tissue metabolism (eg., creatine monohydrate, chromium picolinate, amino acid/protein supplements, beta-hydroxy-beta-methyl-butyrate, anabolic-androgenic steroids, medium- or long-chain fatty acids, branched chain amino acid supplements, amino acids that potentially increase insulin or GH secretion (eg., arginine)) within 1 month of enrollment. These supplements will not be permitted during the treatment period.
21. Dementia or reduced cognitive function or unable to provide voluntary informed consent. Prisoners will not be enrolled.
22. Active substance abuse (e.g., alcoholism, cocaine, heroin, crack, methamphetamine, phencyclidine). Upon evaluation, if the physician-investigator considers that this substance abuse does not put the volunteer at risk for an adverse (ie. cardiovascular) event, or if the physician-investigator feels that the volunteer will be reliable and compliant with the treatment regimens, and that this substance abuse will not interfere with the study medications, exercise regimens, or data interpretation, then at the physician-investigators discretion the volunteer may be eligible.
23. Any cytokine or anti-cytokine therapy during the 3 months prior to enrollment.
24. Patients felt by the Physician Investigator to have uncontrolled hypertension or other diseases (i.e. vasculitis, pulmonary HTN) that otherwise may be a cause of significant underlying or variable endothelial dysfunction
25. Receiving vasoactive substances (i.e. nitrates, viagra) other than antihypertensives that cannot be discontinued at least 12 hours before endothelial function testing (BART).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Reeds DN, Cade WT, Mondy K, Bopp C, Lassa-Claxton S, Yarasheski KE. Pioglitazone ± exercise training reduces liver lipid content and improves insulin sensitivity in HIV with impaired glucose tolerance (IGT). Antivir Ther. 12 Suppl 2: L14, 2007.
- [Result] Yarasheski KE, Cade WT, Overton ET, Mondy KE, Hubert S, Laciny E, Bopp C, Lassa-Claxton S, Reeds DN. Exercise training augments the peripheral insulin-sensitizing effects of pioglitazone in HIV-infected adults with insulin resistance and central adiposity. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E243-51. doi: 10.1152/ajpendo.00468.2010. Epub 2010 Oct 19. PMID 20959530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-infected men and women (18 - 60 yr old) were recruited from the AIDS Clinical Trials Unit, the Infectious Diseases Clinic, and the Volunteers for Health Program at Washington University School of Medicine, St. Louis MO between Jan 2005-Dec 2010. Participants were randomly assigned (1:1) to 4 mo of pioglitazone with or without exercise training.
Pre-assignment Details: Exclusion: AIDS diagnosis, non-compliant with anti-HIV medications, unstable CD4+ T-cell count or plasma HIV viremia, illegal drug abuse.
Period: Overall Study
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Started | 22 | 22
Completed | 20 | 19
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (2) | 46 (2) | 45 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Insulin-stimulated Glucose Disposal Rate
Description: Insulin-mediated glucose disposal rate per kg of fat free mass per min
Time Frame: Baseline and week16
Measure: Mean (Standard Error); unit: µmol glucose/kg FFM/min
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
µmol glucose/kg FFM/min
  Baseline | 30 (4) | 34 (4)
  Week 16 | 37 (6) | 48 (6)

2. Secondary Outcome: Visceral Fat Volume
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: cm3
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
cm3
  Baseline | 1933 (150) | 1890 (217)
  Week 16 | 1970 (164) | 1746 (177)

3. Secondary Outcome: Abdominal Subcutaneous Fat Volume
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: cm3
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
cm3
  Baseline | 2101 (293) | 1877 (197)
  Week 16 | 2164 (286) | 1905 (230)

4. Secondary Outcome: Hepatic Lipid Content
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: percent of water
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
percent of water
  Baseline | 12.1 (2.0) | 8.0 (1.7)
  Week 16 | 10.7 (2.4) | 5.5 (0.8)

5. Secondary Outcome: Hepatic Glucose Production Rate
Description: ability of insulin to suppress hepatic glucose production = hepatic insulin sensitivity
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: percent suppression
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
percent suppression
  Baseline | 32 (3) | 37 (5)
  Week 16 | 40 (6) | 42 (7)

6. Secondary Outcome: Serum Lipid and Lipoprotein Levels
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: mM/L
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
mM/L
  Baseline Triglycerides | 2.3 (0.3) | 2.1 (0.4)
  Week 16 Triglycerides | 2.5 (0.3) | 1.8 (0.2)
  Baseline Total Cholesterol | 4.9 (0.2) | 4.7 (0.2)
  Week 16 Total cholesterol | 4.6 (0.2) | 4.5 (0.2)
  Baseline LDL cholesterol | 2.8 (0.2) | 2.7 (0.2)
  Week 16 LDL cholesterol | 2.5 (0.1) | 2.6 (0.2)
  Baseline HDL cholesterol | 0.99 (0.05) | 1.06 (0.05)
  Week 16 HDL cholesterol | 0.98 (0.05) | 1.09 (0.05)

7. Secondary Outcome: Liver Enzyme Levels
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
U/L
  Baseline ALT | 38 (7) | 34 (6)
  Week 16 ALT | 39 (8) | 32 (6)
  Baseline AST | 34 (7) | 27 (4)
  Week 16 AST | 30 (4) | 27 (3)

8. Secondary Outcome: Hemoglobin
Time Frame: Baseline and Week 16
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
g/L
  Baseline Hemoglobin | 13.8 (0.3) | 13.8 (0.5)
  Week 16 Hemoglobin | 13.7 (0.3) | 13.6 (0.4)

9. Secondary Outcome: Hematocrit
Description: Percentage of blood volume that is red cells
Time Frame: Baseline and Week 16
Measure: Mean (Standard Error); unit: % red cells
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
% red cells
  Baseline Hematocrit | 39.9 (0.7) | 40.7 (1.4)
  Week 16 Hematocrit | 39.6 (0.7) | 39.7 (1.3)

10. Secondary Outcome: Serum Adiponectin Levels
Time Frame: Baseline and week 16
Measure: Mean (Standard Error); unit: µg/mL
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 20 | 19
µg/mL
  Baseline serum adiponectin | 4.7 (0.8) | 4.8 (0.8)
  Week 16 serum adiponectin | 7.0 (0.7) | 6.5 (0.9)

11. Secondary Outcome: Myocardial Contractility
Description: E/A ratio; ratio of the early (E) to late (A) ventricular filling velocities
Time Frame: Baseline and week 16
Population: Number of participants for measures of myocardial contractility is less than that for all other measures. These measures were added to the protocol (after ~50% enrollment) after some reports suggested that this drug class (thiazolidinediones) may adversely affect heart function.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 11 | 10
ratio
  Baseline E/A ratio | 1.3 (0.2) | 1.2 (0.1)
  Week 16 E/A ratio | 1.4 (0.2) | 1.4 (0.1)

12. Secondary Outcome: Myocardial Contractility-LV Ejection Time
Description: Time required to empty the left ventricle into the aorta
Time Frame: Baseline and week 16
Population: as for outcome 11
Measure: Mean (Standard Error); unit: msec
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 11 | 10
msec
  Baseline LV ejection time | 296 (8) | 281 (12)
  Week 16 LV ejection time | 294 (9) | 305 (9)

13. Secondary Outcome: Myocardial Contractility-DT
Description: Deceleration time; time from the peak of early diastolic filling to baseline
Time Frame: Baseline and week 16
Population: as for outcome 11
Measure: Mean (Standard Error); unit: msec
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 11 | 10
msec
  Baseline DT | 204 (7) | 214 (12)
  Week 16 DT | 193 (6) | 190 (4)

14. Secondary Outcome: Myocardial Contractility-SBP
Description: Systolic blood pressure; peak vascular pressure during ventricular contraction
Time Frame: Baseline and week 16
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 11 | 10
mmHg
  Baseline SBP | 114 (2) | 121 (4)
  Week 16 SBP | 114 (2) | 114 (3)

15. Secondary Outcome: Myocardial Contractility-DBP
Description: Diastolic blood pressure; vascular pressure during ventricular relaxation (diastole)
Time Frame: Baseline and week 16
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Number analyzed (Participants) | 11 | 10
mmHg
  Baseline DBP | 65 (3) | 68 (5)
  Week 16 DBP | 67 (4) | 61 (4)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Pioglitazone + Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
No intervention and exercise training only control groups were not included. Intracellular mechanisms were not explored. Relatively small number of participants taking a variety of anti-HIV medication regimens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No